CLINICAL TRIAL: NCT01016795
Title: A Randomized Study of Peripheral Blood Progenitor Cell Priming Comparing a Combination of r-metHuSCF and Filgrastim or Chemotherapy and Filgrastim on Mobilization and Engraftment in Patients With Relapsed or Refractory Lymphomas
Brief Title: Stem Cell Factor (SCF) Priming of Haematopoietic Stem Cell Grafts in Malignant Lymphoma
Acronym: SCF980266
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed Nov 2000 by Amgen, who stopped drug delivery
Sponsor: Aalborg University Hospital (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); University Hospital, Linkoeping (Other); Umeå University (Other); Oslo University Hospital (Other); Nordic Lymphoma Group (Network); Amgen (Industry)
Responsible Party: Hans Erik Johnsen MD DMSc, Professor Clinical Haematology, Department of Haematology Aalborg Hospital Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCF 980266; H-KA-99040-GMS (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2009-11

CONDITIONS: Malignant Lymphoma
Keywords: SCF; Priming; Mobilization; Lymphoma; Clinical Trial
MeSH Terms: conditions — Lymphoma | interventions — ancestim; Filgrastim; Stem Cell Factor; Granulocyte Colony-Stimulating Factor; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- r-metHuSCF and Filgrastim (Active Comparator): Patients were randomized in a 1:1 ratio to either chemotherapy combined with 10 µg/kg/d Filgrastim (control arm B), administered by subcutaneous injection for 14 days, or the combination of 10 µg/kg/d Filgrastim and SCF administered subcutaneously at a dose of 20 µg/kg/d (experimental arm A) for 8 days. Different injection sites were used for each cytokine.
  Interventions: Drug: r-metHuSCF and Filgrastim; Drug: Chemotherapy plus Filgrastim
- Cyclophosphamide and Filgrastim (Active Comparator): Patients were randomized in a 1:1 ratio to either chemotherapy combined with 10 µg/kg/d Filgrastim (control arm B), administered by subcutaneous injection for 14 days, or the combination of 10 µg/kg/d Filgrastim and SCF administered subcutaneously at a dose of 20 µg/kg/d (experimental arm A) for 8 days. Different injection sites were used for each cytokine.
  Interventions: Drug: r-metHuSCF and Filgrastim; Drug: Chemotherapy plus Filgrastim

INTERVENTIONS:
Drug: r-metHuSCF and Filgrastim — Patients were randomized in a 1:1 ratio to either chemotherapy combined with 10 µg/kg/d Filgrastim (control arm B), administered by subcutaneous injection for 14 days, or the combination of 10 µg/kg/d Filgrastim and SCF administered subcutaneously at a dose of 20 µg/kg/d (experimental arm A) for 8 days. Different injection sites were used for each cytokine.
  Other Names: Stem Cell Factor and G-CSF
Drug: r-metHuSCF and Filgrastim — Patients were randomized in a 1:1 ratio to either chemotherapy combined with 10 µg/kg/d Filgrastim (control arm B), administered by subcutaneous injection for 14 days, or the combination of 10 µg/kg/d Filgrastim and SCF administered subcutaneously at a dose of 20 µg/kg/d (experimental arm A) for 8 days. Different injection sites were used for each cytokine.
  Other Names: Stem Cell Factor and G-CSF
  Arms: r-metHuSCF and Filgrastim
Drug: Chemotherapy plus Filgrastim — Patients were randomized in a 1:1 ratio to either chemotherapy combined with 10 µg/kg/d Filgrastim (control arm B), administered by subcutaneous injection for 14 days, or the combination of 10 µg/kg/d Filgrastim and SCF administered subcutaneously at a dose of 20 µg/kg/d (experimental arm A) for 8 days. Different injection sites were used for each cytokine.
  Other Names: Priming chemotherapy and G-CSF

SUMMARY:
Clinical Hypothesis:

It is expected that by removing chemotherapy and adding ancestim to the mobilization scheme in most of the subjects sufficient PBPC will be harvested with a minimum of toxicity and side effects.

DETAILED DESCRIPTION:
Autologous stem cell transplantation is used to support high dose chemotherapy in haematological malignancies.1-2 Peripheral blood progenitor cells (PBPC) have replaced bone marrow cells as the preferred source for transplantation due to faster blood cell recovery.3-4 One variable of major impact for posttransplant care is the number of PBPC harvested.5-8 Therefore, several clinical studies have aimed to identify priming regimens that improve progenitor and stem cell mobilizations and collections without increased toxicity. Frequently, Filgrastim (r-met HuG-CSF) is administrated alone; however, Filgrastim combined with chemotherapy has proven more effective in context of CD34+ cell numbers harvested9-11 and this combination is considered the gold standard for priming and stem cell mobilization in relapsed malignant lymphoma.

Stem cell factor (SCF) is a glycoprotein growth factor that acts on haematopoietic blood cell progenitors.12 Whereas SCF alone exerts little colony-stimulating activity on normal human bone marrow cells in vitro, combination of SCF with other recombinant haematopoietic cytokines results in a synergistic increase in numbers of colonies.13 In vivo, the addition of SCF to G-CSF (Filgrastim) synergistically increases PBPC mobilization compared to Filgrastim alone.14-17 Several clinical trials have reported the ability of the combination of SCF with Filgrastim to mobilize PBPC in patients with lymphoma, multiple myeloma, breast and ovarian cancers even in heavily pretreated patients.18-26 Priming using chemotherapy is toxic and costly11 and new priming procedures need to be established, which is the background for this randomized pilot study. The hypothesis is that elimination of chemotherapy from the priming regimen may decrease the overall toxicity and the ability to collect a sufficient autograft which, however, may be circumvented by adding r-metHuSCF (Ancestim) to the priming regimen. The aim of this randomized phase II trial was to evaluate safety, toxicity and efficacy of growth factors in lymphoma patients considered candidates for high dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Hodgkin's disease and non-Hodgkin lymphomas (Real classification)

  * in relapse
  * refractory to initial chemotherapy
  * with partial response after initial therapy
* Age > 18 years and < 65 years
* ECOG performance status 0, 1 or 2
* Life expectancy of > 6 months with treatment
* ANC > or equal to 1.5 x 109/L, Platelets > or equal to 100 x 109/L
* Serum creatinine < or equal to 150 µmol/L, bilirubin, aspartate aminotransferase (ASAT), and alanine aminotransferase (ALAT) less than twice the upper limit defined at the investigating laboratory
* Prior to mobilization chemotherapy subject has given written informed consent, personally dated

Exclusion Criteria:

* Prior DexaBEAM or miniBEAM therapy and prior bone marrow or PBPC transplant
* Any history of seasonal or recurrent asthma within the preceding 10 years.
* Any history of anaphylactic / anaphylactoid-type event manifested by disseminated urticaria, laryngeal oedema, and / or bronchospasm (example, food, insect bites, etc.). Subjects with drug allergies, manifested solely by rash and / or urticaria, are not excluded
* Any history of angioedema or recurrent urticaria
* Clinical or microbiological evidence of infection at the date of enrollment.
* Subjects with a concurrent malignancy
* Significant non-malignant disease including documented HIV infection, uncontrolled hypertension, unstable angina, congestive heart failure, poorly controlled diabetes, coronary angioplasty within six months, myocardial infarction within the last six months, or uncontrolled atrial or ventricular cardiac arrhythmias
* Pregnant or breast feeding subjects or those of child-bearing potential who are not using adequate contraceptive precautions
* Concurrent enrollment on any other protocol using an investigational drug
* Haematopoietic growth factors administered within one week of study entry
* Subjects with a psychiatric, addictive or any disorder which compromises ability to give truly informed consent for participation in this study
* Known sensitivity to E. coli derived products
* Concurrent use of beta adrenergic blocking agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1999-01; Primary Completion 2000-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and Toxicity was assessed by morbidity, including unexpected adverse events associated with the priming and the transplantation phases during study, and measured and graded by CTC criteria. | From inclusion to 1 months post transplantation

SECONDARY OUTCOMES:
To compare the time dependent level of blood circulating and harvested haematopoietic stem cells and progenitors (PBSC) in patients treated with either a combination of r-metHuSCF and Filgrastim, or conventional chemotherapy plus Filgrastim. | From inclusion to 1 months post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Hans E Johnsen, MD DMSc, Principal Investigator — Aalborg Hospital and Herlev University Hospital
Locations (8):
- Denmark (3):
  - Aalborg Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Copenhagen
- Finland (2):
  - University Hospital Helsinki, Helsinki
  - University Hospital Turku, Turku
- Radiumhospitalet, Oslo, Norway
- Sweden (2):
  - University Hospital Linköping, Linköping
  - University Hospital Umeå, Umeå